CLINICAL TRIAL: NCT04006522
Title: An Exploratory Study of 89Zr-DFO-Atezolizumab ImmunoPET/CT in Patients With Locally Advanced or Metastatic Renal Cell Carcinoma
Brief Title: 89Zr-DFO-Atezolizumab ImmunoPET/CT in Patients With Locally Advanced or Metastatic Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: James Brugarolas (Other)
Responsible Party: Sponsor-Investigator, James Brugarolas, Professor, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STU-2019-0714
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Renal Cell Carcinoma
Keywords: renal cell carcinoma; atezolizumab; PET/CT
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Patients with Localized RCC prior to nephrectomy.
  Interventions: Drug: 89Zr-DFO-Atezolizumab; Procedure: Positron Emission Tomography/Computed Tomography
- Cohort 2 (Experimental): Patients with Unresectable/Metastatic RCC prior to treatment with an immune checkpoint inhibitor.
  Interventions: Drug: 89Zr-DFO-Atezolizumab; Procedure: Positron Emission Tomography/Computed Tomography

INTERVENTIONS:
Drug: 89Zr-DFO-Atezolizumab — 89Zr-DFO-Atezolizumab infusion
Procedure: Positron Emission Tomography/Computed Tomography — PET/CT scan 7 days (± 1 day) after infusion of 89Zr-DFO-Atezolizumab.
  Other Names: PET/CT

SUMMARY:
This is an exploratory clinical trial to assess the potential of 89Zr-DFO-Atezolizumab Positron Emission Tomography/Computed Tomography (PET/CT) scans in patients with locally advanced or metastatic renal cell carcinoma (RCC). This open label, nontherapeutic trial will test the correlation of 89Zr-DFO-Atezolizumab immunoPET/CT with programmed death-ligand 1 (PD-L1) expression and the response to immune checkpoint inhibitor therapy in patients with RCC. There will be two cohorts, one made up of patients with localized RCC who will undergo 89Zr-DFO-Atezolizumab PET/CT prior to nephrectomy and a second cohort of patients with metastatic RCC who will undergo 89Zr-DFO-Atezolizumab PET/CT prior to treatment with an immune checkpoint inhibitor.

DETAILED DESCRIPTION:
PD-L1 expression in tissue of a variety of tumor types has both prognostic and predictive significance for patients treated with immune checkpoint inhibitors. A number of efforts are underway to better identify patients who will benefit from immune checkpoint inhibition. Among these efforts are the use of radiolabeled antibodies against PD-L1. While under investigation in a number of tumor types, to our knowledge this is the first such effort in renal carcinoma, despite the clear evidence of clinical efficacy of immune checkpoint inhibitors in kidney cancer. Our primary aim with this study is to explore 89Zr-DFO-Atezolizumab as a positron emission tomography (PET) tracer in patients with RCC.

The study involves 55 patients distributed across two different groups. The first group is made up of patients with high risk localized disease that will be having surgery. 89Zr-DFO-Atezolizumab PET/CT prior to surgery will be correlated with PD-L1. The second group is made up of patients with unresectable or metastatic RCC that will receive an anti-programmed death 1 (PD1)/programmed death-ligand 1 antibody (alone or in combination). 89Zr-DFO-Atezolizumab PET uptake at site of diseases will be evaluated within and across patients and correlated with treatment responsiveness in exploratory analyses. Patients will be followed for signs of recurrence or progression of their cancer and repeat 89Zr-DFO-Atezolizumab PET scans will be offered at that time. Biopsy after subsequent PET/CT will be strongly encouraged.

Subjects will have data collected during the course of routine clinical care including response to immune checkpoint inhibitor therapy, and toxicities developed during immune checkpoint inhibitor therapy.

This is an exploratory analysis correlating 89Zr-DFO-Atezolizumab uptake with PD-L1 immunohistochemical (IHC) analyses in locally advanced kidney cancer (cohort 1) and will evaluate whether 89Zr-DFO-Atezolizumab uptake across metastatic sites of kidney cancer correlates with known radiographically evident metastatic sites of disease, PD-L1 expression, and response to anti-PD1/PD-L1 immunotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected renal cell carcinoma with planned surgery or patients with metastatic RCC and a tissue diagnosis. (In standard clinical practice, biopsy is not routinely performed in patients who will be having surgery).
* Ability to understand and the willingness to sign a written informed consent.
* Patient must be able to lie still for a 30 to 60 minute PET/CT scan.
* One of the following:

  1. Patients with locally advanced RCC planned for surgery determined to be a high risk of recurrence, defined by presence of at least clinical T2 or TxN1, OR patients with metastatic RCC for whom treatment with cytoreductive nephrectomy and/or metastasectomy is planned by the treating physician.
  2. Patients with metastatic RCC for whom immuno-oncology (IO) therapy is planned.
* Women of child-bearing potential must agree to undergo and have documented a negative pregnancy test on the day of 89Zr-DFO-Atezolizumab administration. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Exclusion Criteria:

* History of severe allergic, anaphylactic, or other hypersensitivity reactions to atezolizumab or any other chimeric or humanized antibodies.
* Uncontrolled severe and irreversible intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
* Significant autoimmune disease requiring treatment with either prednisone (or steroid equivalent) at a dose > 10 mg/day or other immunosuppressive agents. (Replacement steroid therapy is acceptable).
* Any patient for whom ICI therapy would be contraindicated for other reasons. Patients with adverse reactions to ICI therapy may undergo second 89Zr-DFO-Atezolizumab injection and PET/CT at the discretion of the treating physician considering that the dose of antibody represents 1% of a single therapeutic dose and therefore unlikely to cause adverse events.
* Subjects unable to provide informed consent.
* Subjects who are claustrophobic or have other contraindications to PET/CT.
* Subjects must not weigh more than the maximum weight limit for the table for the PET/CT scanner where the study is being performed. (>200 kg or 440 lbs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2019-10-02 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Correlation between 89Zr-DFO-Atezolizumab and PD-L1 | Up to 5 years
  Correlation between 89Zr-DFO-Atezolizumab PET/CT and PD-L1 expression at the time of nephrectomy in patients with localized kidney cancer.
Correlation between 89Zr-DFO-Atezolizumab and anti-PD1/PD-L1 therapy | Up to 5 years
  Correlation between 89Zr-DFO-Atezolizumab PET/CT and response to anti-PD1/PD-L1 therapy.

CONTACTS AND LOCATIONS:
Overall Officials: James Brugarolas, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mulgaonkar A, Elias R, Woolford L, Guan B, Nham K, Kapur P, Christie A, Tcheuyap VT, Singla N, Bowman IA, Stevens C, Hao G, Brugarolas J, Sun X. ImmunoPET Imaging with 89Zr-Labeled Atezolizumab Enables In Vivo Evaluation of PD-L1 in Tumorgraft Models of Renal Cell Carcinoma. Clin Cancer Res. 2022 Nov 14;28(22):4907-4916. doi: 10.1158/1078-0432.CCR-22-1547. PMID 36074149